CLINICAL TRIAL: NCT07082348
Title: Assessing the Feasibility and Potential Efficacy of Herbs and Spices for Improving Dietary Quality and Adherence to the Dietary Guidelines for Americans in College Students With Poor Dietary Quality: A Pilot Study
Brief Title: Feasibility and Potential Efficacy of Herbs and Spices for Improving Dietary Quality in College Students: A Pilot Study
Acronym: HerbSpicesDiet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: McCormick Science Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UNLV-2024-569
Record Dates: First submitted 2025-06-11; First posted 2025-07-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-06

CONDITIONS: Dietary Quality; Feasibility Studies; College Student; Dietary Guidelines for Americans; Gut Microbiome; Lipid Profiles; Herbs and Spices; Acceptability; Inflammation Biomarkers; Body Composition; Anthropometrics
Keywords: dietary quality; dietary guidelines for americans; college students; cardiometabolic health; gut microbiome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Herbs and Spices Nutrition Education Program (Experimental): Participants will attend two group visits at the UNLV Nutrition Center (weeks 0 and 3 of the 6-week intervention), where trained RDs will deliver the HSNP, covering the principles and health benefits of the Dietary Guidelines for Americans (DGA), recommended food group intake, and practical, budget-friendly strategies for incorporating herbs and spices into the diet. Sessions will include education, supporting materials, and a sensory evaluation of 20 foods (spanning fruits, vegetables, grains, dairy, and proteins) prepared with various herbs and spices, rated using a 9-point hedonic scale to identify preferred flavor profiles and promote long-term DGA adherence through enhanced taste and acceptability.
  Interventions: Behavioral: Herbs and Spices Nutrition Education Program

INTERVENTIONS:
Behavioral: Herbs and Spices Nutrition Education Program — Participants will attend two group visits at the UNLV Nutrition Center (weeks 0 and 3 of the 6-week intervention), where trained RDs will deliver the HSNP, covering the principles and health benefits of the Dietary Guidelines for Americans (DGA), recommended food group intake, and practical, budget-friendly strategies for incorporating herbs and spices into the diet. Sessions will include education, supporting materials, and a sensory evaluation of 20 foods (spanning fruits, vegetables, grains, dairy, and proteins) prepared with various herbs and spices, rated using a 9-point hedonic scale to identify preferred flavor profiles and promote long-term DGA adherence through enhanced taste and acceptability.

SUMMARY:
The goal of this single-arm feasibility, pilot study is to assess the feasibility, acceptability, and potential effectiveness of the Herbs and Spices Nutrition Education Program (HSNP-focusing on incorporating herbs and spices into the diet for adherence to the DGA's) for determining the scalability of implementing this intervention for a larger scale, more comprehensive study The main questions it aims to answer are:

* What is the feasibility and acceptability of incorporating herbs and spices into the diet along with DGA-focused nutrition education through the HSNP in college students with poor dietary quality?
* What are the preliminary effects of the HSNP on dietary intake/quality, cardiometabolic, and gut health in college students with poor dietary quality?
* What are the barriers associated with HSNP implementation in college students with poor dietary quality?

Participants will:

* Be asked to come to the study site initially for a Screening Study Visit to confirm eligibility.
* Be asked to come the clinical study site for a Pre-HSNP and Post-HSNP Study Visit (one week prior starting the HSNP and after week 6 of completing the HSNP) for assessments of cardiometabolic and gut health.
* Be asked to come to the Nutrition Center for weeks 0 and 3 of the HSNP, where they will receive education on the Dietary Guidelines for Americans and the health benefits of herbs and spices, have a sensory evaluation of foods, be provided budget-friendly recipes and resources, and given take-home herbs, spices, and supporting materials
* Be asked to complete 3-Day Food Records throughout the 6 week study period for assessment of dietary quality (4 total)

DETAILED DESCRIPTION:
Study Overview: Investigators will recruit 30 college students experiencing poor dietary quality, to participate in this 6-week pilot, single-arm clinical trial. Participants will be recruited from the metropolitan Las Vegas area through campus and community advertisements including flyers, newspaper articles, social media, and public events. Randomization will not be needed as all participants recruited will be receiving the intervention. There will be two cohorts of 15 participants for the 6-week HSNP.

Prescreen Interview: Potential participants who inquire about the study by calling the recruitment phone line or by QR code via Qualtrics, will be given a brief overview of the study and will be asked a series of questions to determine whether they should be invited for the in-person screening visit. Eligibility will be based on inclusion/exclusion criteria and responses to questions about medical history and dietary habits. Potential participants will be invited to report to the clinical facilities in the Bigelow Health Sciences Building at UNLV (study site) for their first on-site visit (and all subsequent study visits if the participant qualifies) to ascertain eligibility (screening study visit). This pre-screening interview will occur prior to participants consenting (which occurs at the in person screening study visit).

Screening Study Visit: Potentially eligible participants will be invited to the Functional Foods and Health Lab (BHS313) of the Rod Lee Bigelow, Health Sciences Building at UNLV (health assessment-study site) for their first on-site visit for screening (and subsequent 2 study visits if the participant qualifies for the future Pre and Post-HSNP Visits) to ascertain eligibility. During this screening study visit, the potential participants will be provided with verbal and written explanations of the project and will have any questions regarding the study answered by trained research personnel during the informed consent process. Consenting participants will be asked to sign an informed consent document (with a copy provided to the participant to take home). Screening will consist of determination of dietary quality using the Global Diet Quality Score, their adherence to dietary guidelines using the Rapid Prime Diet Quality Score Screener, SES Questionnaire, an Herbs and Spices Questionnaire to determine usual herbs and spices intake, and nutrition knowledge using the General Nutrition Knowledge Questionnaires. Anthropometrics and blood pressure will be measured and questions regarding medical history and medication use will be asked during the screening visit to confirm eligibility. Should the results of anthropometrics and/or blood pressure fall outside the range for inclusion, participants will be promptly notified and excluded from further participation before any additional data is collected. If participants meet the inclusion criteria for the study, they will be asked to come for subsequent study visits (Pre- and Post-HSNP Study Visits) and be a part of the 6-week HSNP Program. Participants who are not eligible will be thanked for their time and participation and told the specific reasoning for why they do not meet the inclusion criteria. Eligible participants will be asked to complete a three-day food record using NCI's Automated Self-Administered 24-Hour Dietary Assessment Tool to assess typical dietary intake and dietary quality (Healthy Eating Index [HEI]-2020 scoring), prior to their Pre-HSNP Study Visit at participants homes via a computer, ipad, or smartphone. The Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24) is a web-based dietary recall system developed by the National Cancer Institute. It allows participants to self-report their dietary intake over the past 24 hours using a user-friendly interface that prompts for detailed food and beverage consumption. The tool can be distributed via a unique web link provided to participants, enabling remote data collection without requiring in-person visits.

Fecal Sample Collection for Assessment of Gut Microbiome: After participants confirm eligibility from their screening visit, they will be given a "Fecal Collection Tube" with instructions provided. Participants will be asked to collect a sample in the privacy of your own home, to bring back with them to their Pre-HSNP Study Visit. Participants will prepare and collect a fecal sample using the provided tube. The collection tube cap will be unscrewed, and a small spoon will be provided to scoop one spoonful of feces. The fecal sample will then be placed in the collection tube. Finally, participants will tighten the cap and shake to mix the contents. The sample is fine to be stored at room temperature prior to bringing to BHS313 for the pre and post-HSNP Study Visits. Participants will also receive another Fecal Collection Tube at the end of their HSNP week-3 visit at the Nutrition Center to complete prior to coming in for their Post-HSNP Study visit, following all the same procedures as above.

Pre- and Post-HSNP Study Visit: Participants will be asked to come fasted to the study site (between 7:00-10:00 A.M., 12 hours after the abstinence from caffeine and 24 hours after the last bout of moderate/heavy physical activity); vascular assessments (blood pressure, Pulse Wave Velocity, Pulse Wave Analysis) will be measured followed by body composition (Bioelectrical Impedance Analysis), finger prick blood draw (fasting blood glucose and lipid profiles, venous blood draw (inflammatory and oxidative stress biomarkers), anthropometrics (height, weight, and waist/hip circumference), assessment of fruit and vegetable intake via Raman Spectroscopy, assessment of physical activity patterns (Five-City Project Physical Activity Recall), nutrition knowledge (General Nutrition Knowledge Questionnaire), Mood State (Profile of Mood States Questionnaire), Gastrointestinal Health Questionnaires, and sleep quality (Pittsburg Sleep Quality Index).

Herbs and Spices Nutrition Education Program: Participants will visit the UNLV Nutrition Center for two visits after completion of their Pre-HSNP Study Visit at weeks 0 and 3 of the 6-week intervention to receive the HSNP in a group format (15 participants in each group), which our research team equipped with RD's has had experience creating and leading nutrition and education programs. HSNP will include an explanation of the principles and components of the Dietary Guidelines for Americans (DGA), health benefits of following the DGA, how to incorporate herbs and spices in the diet, guidance on recommended intake of various food groups, budget-friendly strategies and recipes for incorporation of herbs and spices in the diet, and supporting resources such as educational materials and online tools. Participants will then complete a sensory evaluation using the 9-point hedonic scale for 20 foods (including four different recipes for vegetables, fruits, grains/grain products, dairy products, and proteins/protein alternatives) prepared with various herbs and spices.

Dietary Assessments During Weeks 0, 2, 4, and 6 of Intervention Period: Participants will be asked to complete a three-day food record using NCI's Automated Self-Administered 24-Hour (ASA24) Dietary Assessment Tool to assess typical dietary intake and diet quality (using HEI-202075) during weeks 0, 2, 4, and 6 of the intervention period. This food record can be completed at any point during weeks 0, 2, 4, and 6 of intervention the period at participants' homes via a computer or ipad.

ELIGIBILITY:
Inclusion Criteria:

* College students (undergraduate and graduate)
* Ages 18-39 years
* BMI 18.5-40 kg/m
* Having poor dietary quality (a Rapid Prime Diet Quality Score of 12 or below),
* Maintain current lifestyle habits (e.g., medications/ supplement use, exercise, and sleep), and avoid taking new supplements or medications throughout the study.

Exclusion Criteria:

* Individuals diagnosed with myocardial infarction within the past 6 months
* Uncontrolled hypertension
* BMIs <18.5 or >40 kg/m2
* Autoimmune disease or immune compromised
* A recent diagnosis of cancer or under current treatment for cancer
* A history of kidney stones
* Having pacemaker
* Participating in a weight loss program
* Having a history of any significant GI disease
* Insulin use
* Currently on dialysis
* Currently consuming pro-/pre-biotics or antiobiotics
* Diagnosed with unstable chronic metabolic disease
* Have allergies to any herbs and spices
* Are pregnant/nursing
* Participating in another investigational study
* Unable or unwilling to give consent

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Dietary Quality | Pre- and Post- HSNP: 6 weeks
  Dietary Quality measured via Health Eating Index-2020 from three-day food records using NCI's Automated Self-Administered 24-Hour Dietary Assessment Tool. The index score will be from 0-100, with 0 indicating poorest diet quality and 100 excellent.
Changes In Dietary Intake | Pre- and Post- HSNP: 6 weeks
  Dietary intake measured from three-day food records using NCI's Automated Self-Administered 24-Hour Dietary Assessment Tool, will be measured throughout the study period to indicate any changes in overall macro and micro nutrient intake between the treatment and comparative control group.
Feasibility of HSNP | Pre- and Post- HSNP: 6 weeks
  To recruit at least 80% of the target sample size (24 out of 30 participants), retain at least 85% of enrolled participants through to the end HSNP (no more than 4 dropouts), deliver ≥90% of planned HSNP intervention, and collect ≥90% of three-day food records through the study period.
Adherence of HSNP | Pre- and Post- HSNP: 6 weeks
  To have ≥80% of participants completing the whole HSNP (attending both study visits and nutrition education sessions; 24 out of 30 participants)
Acceptability of HSNP | Pre- and Post- HSNP: 6 weeks
  To asses acceptability at the 3-week HSNP visit and upon completing of HSNP via survey and optional semi-structured interviews. The survey will include Likert-Scale items (1-5 and 1-10) across satisfaction, perceived relevance, taste, convenience, and likelihood of continued use.

SECONDARY OUTCOMES:
Change in Fasting Blood Glucose Levels | Pre- and Post- HSNP: 6 weeks
  Fasting Blood Glucose Levels Measured with a Glucometer
Change in Lipid Profiles | Pre- and Post-HSNP: 6 weeks
  Measure of fasted lipid profiles (total cholesterol, triglycerides, high-density lipoprotein-cholesterol, low-density lipoprotein-cholesterol) all measured in milligrams per deciliter (mg/dL) via Cholestech LDX Analyzer
Change in Blood Pressure | Pre- and Post-HSNP: 6 weeks
  Fasted diastolic and systolic blood pressure, measured via OMRON automated blood pressure device
Changes in Arterial Stiffness-Pulse Wave Velocity | Pre- and Post-HSNP: 6 weeks
  Fasted measured of arterial stiffness via carotid-femoral and aortic pulse wave velocity (cfPWV) in meters per second (m/s) (SphygmoCor XCEL).
Changes in Arterial Stiffness-Augmentation Index | Pre- and Post-HSNP: 6 weeks
  Fasted measured of arterial stiffness via pulse wave analysis (SphygmoCor XCEL) with measure of Augmentation Index (AIx) expressed as a percentage (%)
Changes in Arterial Stiffness- Central Systolic Blood Pressure | Pre- and Post- HSNP: 6 weeks
  Fasted measured of Central Systolic Blood Pressure (cSBP) measured in mmHg (millimeters of mercury) via SphygmoCor XCEL.
Changes in Arterial Stiffness-Central Pulse Pressure | Pre- and Post-HSNP: 6 weeks
  Fasted measured of Central Pulse Pressure measured in mmHg (millimeters of mercury) via SphygmoCor XCEL.
Changes in Arterial Stiffness-Augmented Pressure | Pre- and Post-HSNP: 6 weeks
  Fasted measured of Augmented Pressure measured in mmHg (millimeters of mercury) via SphygmoCor XCEL
Changes in Arterial Stiffness-Subendocardial Viability Ratio | Pre- and Post- HSNP: 6 weeks
  Fasted measured of arterial stiffness via pulse wave analysis (SphygmoCor XCEL) with measure of Subendocardial Viability Ratio expressed as a percentage (%)
Changes In Arterial Stiffness-Transit Time | Pre- and Post-HSNP: 6 weeks
  Fasted measured of arterial stiffness via transit in milliseconds (SphygmoCor XCEL)
Changes in waist and hip circumferences | Pre- and Post- HSNP: 6 weeks
  Waist and hip circumference changes measured in centimeters.
Change in body fat % | Pre- and Post- HSNP: 6 weeks
  Body fat % measured via Bioelectrical Impedance Analysis (Seca BIA Platform mBCA 554 Medical Body Composition Analyzer)
Changes in Nutrition Knowledge | Pre- and Post- HSNP: 6 weeks
  Measurements of nutrition knowledge via General Nutrition Knowledge Questionnaire which are general questions used to assess a person's understanding of basic nutrition principles and dietary guidelines.
Changes in Fruit and Vegetable Intake Adherence | Pre- and Post HSNP: 6 weeks
  Assessment of fruit and vegetable intake will be measured via Raman Spectroscopy (VeggieMeter)
Changes in Physical Activity Patterns | Pre- and Post- HSNP: 6 weeks
  Assessment of physical activity patterns via Five-City Project Physical Activity Recal
Changes in Sleep Quality | Pre- and Post- HSNP: 6 weeks
  Assessment of sleep quality measured via Pittsburg Sleep Quality Index wich is a questionnaire used to assess the quality and patterns of sleep over a one-month period, measuring factors like sleep duration, sleep disturbances, and daytime dysfunction. The scores are typically presented as a global score, ranging from 0 to 21, where higher scores indicate poorer sleep quality.
Changes in body weight | Pre- and Post- HSNP: 6 weeks
  Body weight will be measured in kilograms with a weighing scale
Changes in Body Mass Index | Pre- and Post- HSNP: 6 weeks
  Body Mass Index will be assessed with a participants height in meters and body weight in kilograms, in the unit of kg/m2
Assessment of Height | Screening
  Height will be assessed in meters (for assessment of BMI at future visits and inclusion criteria)
Changes in High Sensitive C-Reactive Protein | Pre- and Post- HSNP: 6 weeks
  Fasted measure of plasma high sensitivity C-Reactive Protein in mg/L measured via ELISA
Changes in Interleukin-6 | Pre- and Post-HSNP: 6 weeks
  Fasted measure of plasma Interleukin-6 in pg/mL measured via ELISA
Change in Oxidized-LDL | Pre- and Post-HSNP: 6 weeks
  Fasted plasma oxidized LDL (U/L) will be measured via ELISA
Change in Lipopolysaccharide Binding Protein | Pre- and Post- HSNP: 6 weeks
  Fasted measure of plasma Lipopolysaccharide Binding Protein in ng/mL measured via ELISA
Changes in Gut Microbiome | Pre- and Post- HSNP: 6 weeks
  Fecal sample collection of Alpha and Beta Diversity from 16S rRNA
Changes in Gastrointestinal Health | Pre- and Post- HSNP: 6 weeks
  To measure the presence, frequency, history and severity of digestive symptoms such as bloating, gas, abdominal pain, diarrhea, constipation, and overall gut discomfort.
Changes in Mood (Profile of Mood States Questionnaire) | Pre- and Post- HSNP: 6 weeks
  Measure of an individuals current mood across several emotional states, including tension, depression, anger, fatigue, confusion, and vigor.

CONTACTS AND LOCATIONS:
Overall Officials: Neda S Akhavan, PhD, RD, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- Department of Kinesiology and Nutrition Sciences, Las Vegas, Nevada, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared because the study did not obtain participant consent for data sharing, and there are concerns regarding the protection of participant privacy and confidentiality. Additionally, institutional and regulatory policies restrict data sharing, and the data are not intended for broader dissemination.